CLINICAL TRIAL: NCT04791345
Title: Study of the Excretion of Orally Administered Corticosteroids for the Improval of the Detection of Said Substances in Anti-doping Controls
Acronym: DACORSIN/4
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IMIMFTCL/DACORSIN/4
Record Dates: First submitted 2021-03-05; First posted 2021-03-10 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Healthy Volunteers
Keywords: Anti-doping control; Glucocorticoids; Corticosteroids; Dexamethasone; Methylprednisolone; Deflazacort
MeSH Terms: interventions — Methylprednisolone; deflazacort; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Single-center, non-randomized, open-label clinical trial in healthy male volunteers. A single dose of DEX, MP and DEF, and multiple dose of DEX and MP will be administered to different subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Methylprednisone single-dose (Experimental): Subjects receive a single dose treatment. Urine samples will be collected until 5 days after administration in 10 fractions: 0-4h, 4-8h, 8-12h, 12-24h, 24-36h, 36-48h, 48-72h, 72-96h, 96-120h post-administration. Blood samples will be collected until 6 days after administration in 5 fractions: pre-administration and 24h, 48h, 72h and 120h post-administration.
  Interventions: Drug: Methylprednisone
- Methylprednisone multiple-dose (Experimental): Subjects receive a multiple dose treatment. Urine samples will be collected until 7 days after administration in 20 fractions.
  Interventions: Drug: Methylprednisone
- Deflazacort single-dose (Experimental): Subjects receive a single-dose treatment. Urine samples will be collected until 5 days after administration in 10 fractions: 0-4h, 4-8h, 8-12h, 12-24h, 24-36h, 36-48h, 48-72h, 72-96h, 96-120h post-administration. Blood samples will be collected until 6 days after administration in 5 fractions: pre-administration and 24h, 48h, 72h and 120h post-administration.
  Interventions: Drug: Deflazacort
- Dexamethasone single-dose (Experimental): Subjects receive a single-dose treatment. Urine samples will be collected until 13 days after administration in 11 fractions: 0-4h, 4-8h, 8-12h, 12-24h, 24-36h, 36-48h, 48-72h, 72-96h, 96-120h, 120-144h post-administration.
  Blood samples will be collected until 9 days after administration in 6 fractions: pre-administration and 24h, 48h, 72h, 120h and 192h post-administration.
  Interventions: Drug: Dexamethasone
- Dexamethasone multiple-dose (Experimental): Subjects receive a multiple dose treatment. Urine samples will be collected until 10 days after administration in 34 fractions. Blood samples will be collected until 13 days after the first administration.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Methylprednisone — 12 mg of methylprednisone (3 pills of 4 mg each) administered orally in a single dose.
  Other Names: Urbason®
  Arms: Methylprednisone single-dose
Drug: Methylprednisone — 12 mg of methylprednisone (3 pills of 4 mg each) administered orally every 24 hours during 3 days.
  Other Names: Urbason®
  Arms: Methylprednisone multiple-dose
Drug: Deflazacort — 30 mg of deflazacort (1 pill) administered orally in a single dose.
  Arms: Deflazacort single-dose
Drug: Dexamethasone — 4 mg of dexamethasone (1 pill) administered orally in a single dose.
  Arms: Dexamethasone single-dose
Drug: Dexamethasone — 2 mg of dexamethasone (1/2 pill) administered orally every 12 hours during 5 days.
  Arms: Dexamethasone multiple-dose

SUMMARY:
Background:

Glucocorticoids (GC) were included in the list of banned substances in sports in 1986, because of evidences of positive effects on physical performance and the important health risks associated with its consumption.

Due to the fact that GC are commercialized in a variety of pharmaceutical forms and are administered in different ways, it is necessary to establish discrimination criteria to guarantee the therapeutic use of these drugs and to prevent doping.

Hypothesis:

Discrimination criteria between allowed and prohibited administrations of GC must be specific for each of the compounds. Further studies are needed to provide discrimination criteria related to oral administration of GC.

Objectives:

To conduct excretion studies with dexamethasone, methylprednisolone and deflazacort in order to define notification levels and wash-out periods after the administration of a single dose (DEX, MP and DEF) or repeated doses (DEX and MP) of these drugs.

Methods:

Non-randomized, open-label, pharmacokinetics clinical trial where a single dose of DEF, MP and DEX and also a multi-dose of DEX and MP will be administered orally to healthy volunteers (total n=50).

DETAILED DESCRIPTION:
The World Anti-Doping Agency (WADA) has established a general notification level of 30 ng/mL for GC to discriminate allowed and not allowed administrations. However, recent studies have proven that the use of a unique criteria is not adequate given the diversity of administration routes, doses and pharmacokinetics and pharmacodynamics properties of each drug.

The goal of this study is to conduct additional studies using dexamethasone (DEX), methylprednisolone (MP) and deflazacort (DEF) in order to generate additional data of urinary concentrations and wash-out periods after single and repeated oral doses of these drugs.

ELIGIBILITY:
Inclusion Criteria:

* Male volunteers aged between 18 and 55 years.
* Able to understand and accept the trial procedures and able to sign an informed consent prior to any study-mandated procedure.
* History and physical examination that demonstrate not presenting organic or psychiatric disorders.
* ECG, blood and urine tests performed before the experimental session within normal limits. Minor or occasional variations of these limits will be allowed if, in the opinion of the Principal Investigator and taking into account the state of science, they have no clinical significance, do not pose a risk to the subject and do not interfere in the product evaluation. These variations and their non-relevance will be specifically justified in writing.
* Body mass index (weight/height^2) between 19 and 27 kg/m2 and weight between 50 and 100 kg. BMI of 27-28 kg/m2 may be included according to Principal Investigator's criteria.

Exclusion Criteria:

* Failure to meet inclusion criteria.
* History of allergy, idiosyncrasy, hypersensitivity or adverse reactions to glucocorticoids or any of the excipients. Serious adverse reactions to any drug.
* Contraindications to treatment with study drugs (according to the respective summary of product characteristics, SmPC).
* Clinical background or evidence of gastrointestinal, hepatic, renal disorder or others that may involve an alteration of the absorption, distribution, metabolism or excretion of the drug.
* Clinical background or evidence of psychiatric disorders, alcoholism, drug abuse or habitual consumption of psychoactive drugs.
* Having participated in another clinical trial with medication in the three months prior to the start of the study.
* Having donated blood in the three months prior to the start of the study, in the event that blood extractions are made.
* Having suffered some organic disease or major surgery in the six months prior to the start of the study.
* Clinical background or evidence of cardiovascular, respiratory, renal, hepatic, endocrine, gastrointestinal, hematological, neurological, or other acute or chronic diseases that, in the opinion of the Principal Investigator or the collaborators designated by him/her, may pose a risk to the subjects or may interfere with the objectives of the study. Especially osteoporosis, hypertension, Cushing syndrome, diabetes mellitus, and viral infections such as herpes or varicella.
* Having taken medication regularly in the month prior to the study sessions -in case of glucocorticoids 3 months prior- with the exception of vitamins, herbal remedies or dietary supplements that, in the opinion of the Principal Investigator or the collaborators designated by him/her, may not pose a risk to the subjects or may not interfere with the objectives of the study. Treatment with a single dose of symptomatic medication in the week prior to the study sessions will not be a reason for exclusion if it is assumed that the drug has been completely eliminated on the day of the experimental session.
* Smokers of more than 20 cigarettes a day in the 3 months before the study.
* Consumption of more than 40 g of alcohol daily.
* Consumers of more than 5 coffees, teas, cola drinks, or other stimulant drinks or with xanthines daily in the 3 months prior to the study start.
* Being unable to understand the nature, consequences of the trial and the procedures that are asked to follow.
* Positive serology for hepatitis B, C or HIV.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-02-26 (Actual); Primary Completion 2022-02-26 (Estimated); Study Completion 2022-02-26 (Estimated)

PRIMARY OUTCOMES:
Urine concentration of methylprednisone | 0-4h (hours), 4-8h, 8-12h, 12-24h, 24-36h, 36-48h, 48-72h, 72-96h, 96-120h post-administration
  Concentration of methylprednisone in each fraction of urine samples
Urine concentration of methylprednisone metabolites | 0-4h (hours), 4-8h, 8-12h, 12-24h, 24-36h, 36-48h, 48-72h, 72-96h, 96-120h post-administration
  Concentration of methylprednisone metabolites in each fraction of urine samples
Urine concentrations of deflazacort | 0-4h (hours), 4-8h, 8-12h, 12-24h, 24-36h, 36-48h, 48-72h, 72-96h, 96-120h post-administration
  Concentration of deflazacort in each fraction of urine samples
Urine concentrations of deflazacort metabolites | 0-4h (hours), 4-8h, 8-12h, 12-24h, 24-36h, 36-48h, 48-72h, 72-96h, 96-120h post-administration
  Concentration of deflazacort metabolites in each fraction of urine samples
Urine concentration of dexamethasone | 0-4h (hours), 4-8h, 8-12h, 12-24h, 24-36h, 36-48h, 48-72h, 72-96h, 96-120h, 120-144h post-administration
  Concentration of dexamethasone in each fraction of urine samples
Urine concentration of dexamethasone metabolites | 0-4h (hours), 4-8h, 8-12h, 12-24h, 24-36h, 36-48h, 48-72h, 72-96h, 96-120h, 120-144h post-administration
  Concentration of dexamethasone metabolites in each fraction of urine samples

SECONDARY OUTCOMES:
Plasma concentrations of drug metabolites | Before drug administration and at 0.5h (hours), 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 24h, 48h, 72h, 120h, 192h post-administration
  Concentrations of drug metabolites (DEX, MP, DEF) in plasma
Plasma concentrations of cortisol | Before drug administration and at 0.5h (hours), 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 24h, 48h, 72h, 120h, 192h post-administration
  Concentrations of cortisol in plasma
Plasma concentrations of endogen steroids | Before drug administration and at 0.5h (hours), 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 24h, 48h, 72h, 120h, 192h post-administration
  Concentrations of endogen steroids in plasma [testosterone (T), epitestosterone (E), androsterone (A), etiocholanolone (Etio), 5α-androstane-3α,17β-diol (5aAdiol), 5β-androstane-3α,17β-diol (5bAdiol), and the quotients T/E, A/T, A/Etio, 5aAdiol/5bAdiol and 5aAdiol/ET]
Plasma concentrations of testosterone | Before drug administration and at 0.5h (hours), 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 24h, 48h, 72h, 120h, 192h post-administration
  Concentrations of testosterone in plasma
Plasma concentrations of epitestosterone | Before drug administration and at 0.5h (hours), 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 24h, 48h, 72h, 120h, 192h post-administration
  Concentrations of epitestosterone in plasma
Plasma concentrations of androsterone | Before drug administration and at 0.5h (hours), 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 24h, 48h, 72h, 120h, 192h post-administration
  Concentrations of androsterone in plasma
Plasma concentrations of etiocholanolone | Before drug administration and at 0.5h (hours), 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 24h, 48h, 72h, 120h, 192h post-administration
  Concentrations of etiocholanolone (Etio) in plasma
Plasma concentrations of 5α-androstane-3α,17β-diol | Before drug administration and at 0.5h (hours), 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 24h, 48h, 72h, 120h, 192h post-administration
  Concentrations of 5α-androstane-3α,17β-diol (5aAdiol) in plasma
Plasma concentrations of 5β-androstane-3α,17β-diol | Before drug administration and at 0.5h (hours), 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 24h, 48h, 72h, 120h, 192h post-administration
  Concentrations of 5β-androstane-3α,17β-diol (5bAdiol) in plasma
Quotient testosterone/epitestosterone in plasma | Before drug administration and at 0.5h (hours), 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 24h, 48h, 72h, 120h, 192h post-administration
  Concentrations of testosterone/epitestosterone (T/E) in plasma
Quotient androsterone/testosterone in plasma | Before drug administration and at 0.5h (hours), 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 24h, 48h, 72h, 120h, 192h post-administration
  Concentrations of androsterone/testosterone (A/T) in plasma
Quotient androsterone/Etio in plasma | Before drug administration and at 0.5h (hours), 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 24h, 48h, 72h, 120h, 192h post-administration
  Concentrations of androsterone/etiocholanolone (A/Etio) in plasma
Quotient 5aAdiol/5bAdiol in plasma | Before drug administration and at 0.5h (hours), 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 24h, 48h, 72h, 120h, 192h post-administration
  Concentrations of 5α-androstane-3α,17β-diol/5β-androstane-3α,17β-diol (5aAdiol/5bAdiol) in plasma
Quotient 5aAdiol/ET in plasma | Before drug administration and at 0.5h (hours), 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 24h, 48h, 72h, 120h, 192h post-administration
  Concentrations of 5α-androstane-3α,17β-diol/etiocholanolone (5aAdiol/ET) in plasma
Hemoglobin concentration | At -72h (hours), -48h, -24h (before first administration), and at 0h, 1h, 3h, 6h after each dose (in multiple-dose treatments)
  Variation of hemoglobin concentrations in blood
Hematocrit | At -72h (hours), -48h, -24h (before first administration), and at 0h, 1h, 3h, 6h after each dose (in multiple-dose treatments)
  Variation of hematocrit value in blood
Mean corpuscular hemoglobin | At -72h (hours), -48h, -24h (before first administration), and at 0h, 1h, 3h, 6h after each dose (in multiple-dose treatments)
  Variation of mean corpuscular hemoglobin (MCH) levels in blood
Mean corpuscular volume of erythrocytes | At -72h (hours), -48h, -24h (before first administration), and at 0h, 1h, 3h, 6h after each dose (in multiple-dose treatments)
  Variation of mean corpuscular volume of erythrocytes (MCV) levels in blood
Erythrocytes count | At -72h (hours), -48h, -24h (before first administration), and at 0h, 1h, 3h, 6h after each dose (in multiple-dose treatments)
  Variation of erythrocytes count in blood
Standard deviation of the range of distribution of erythrocytes | At -72h (hours), -48h, -24h (before first administration), and at 0h, 1h, 3h, 6h after each dose (in multiple-dose treatments)
  Variation of standard deviation of the range of distribution of erythrocytes
Platelet count | At -72h (hours), -48h, -24h (before first administration), and at 0h, 1h, 3h, 6h after each dose (in multiple-dose treatments)
  Variation of platelet count in blood
Reticulocyte count | At -72h (hours), -48h, -24h (before first administration), and at 0h, 1h, 3h, 6h after each dose (in multiple-dose treatments)
  Variation of reticulocyte count in blood
Fraction of immature reticulocytes | At -72h (hours), -48h, -24h (before first administration), and at 0h, 1h, 3h, 6h after each dose (in multiple-dose treatments)
  Variation of immature reticulocytes fraction in blood

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Ventura Alemany, PharmD, PhD, Principal Investigator — IMIM (Hospital del Mar Medical Research Institute); Ana M Aldea Perona, MD, PhD, Principal Investigator — IMIM (Hospital del Mar Medical Research Institute)
Locations (1):
- IMIM (Hospital del Mar Medical Research Institute), Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No